CLINICAL TRIAL: NCT03783988
Title: An Open, Uncontrolled Pharmacokinetic Study With a New Topical Combination Gel Containing Triiodothyroacetic Acid (TRIAC) and Dehydroepiandrosterone (DHEA) in Subjects With Skin Atrophy Due to Topical Treatment With Glucocorticoids
Brief Title: Study With a Topical Gel Containing TRIAC and DHEA in Subjects With Skin Atrophy Due to Glucocorticoids
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trophea Development AB (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRO-SA01
Record Dates: First submitted 2018-12-03; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Skin Atrophy
MeSH Terms: interventions — Dehydroepiandrosterone; 3,3',5-triiodothyroacetic acid

STUDY DESIGN:
Intervention Model Description: This is a pharmacokinetic study to study the systemic levels of DHEA, DHEAs and TRIAC, before and after application of a new topical combination gel containing DHEA and TRIAC. MS-based validated methods will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open uncontrolled pharmacokinetic study (Other): Single armed - All subjects receive one dose of topical combination gel containing TRIAC and DHEA
  Interventions: Combination Product: DHEA and TRIAC

INTERVENTIONS:
Combination Product: DHEA and TRIAC — The new topical gel contains dehydroepiandrosterone (DHEA) and triiodothyroacetic acid (TRIAC)

SUMMARY:
An open, uncontrolled pharmacokinetic study with a new topical combination gel containing triiodothyroacetic acid (TRIAC) and dehydroepiandrosterone (DHEA) in subjects with skin atrophy due to topical treatment with glucocorticoids.

DETAILED DESCRIPTION:
At the Baseline Visit (Day 1) and after completion of all evaluations, each subject who qualifies for entry will will receive a dose of 0.5 g IMP on the back of a hand affected with skin atrophy.

PK-samples will be withdrawn at 0, 2, 4, 6, 24, 48 and 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained prior to initiating any study specific procedures
2. Men and women of at least 18 years old
3. Subjects with hand eczema and confirmed skin atrophy on the back of a hand caused by treatment with topical glucocorticoids for at least 6 months
4. Atrophic skin area of approximately 100 cm2 (back of a hand)
5. Females of childbearing potential must have a negative urine pregnancy test result upon entry into the study
6. Females of child-bearing potential may participate only if using reliable means of contraception

Exclusion Criteria:

1. Skin atrophy with open ulcer(s) involved
2. Participation in any other study involving investigational drug(s) within 30 days prior to study entry
3. Use of systemic or topical glucocorticoids, thyroid hormones, vitamin A analogues, DHEA, and testosterone within 3 weeks before entry into the study
4. Known thyroid disease of any type
5. Women with polycystic ovary syndrome (PCO), congenital adrenal hyperplasia or other androgen excess syndromes
6. Subjects who have previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in systemic levels (ng/ml) of DHEA after a single topical administration, from baseline (hours) to 72 hours. | 0-72 hours
  MS-based method for analysis of DHEA will be used.
Change in systemic levels (ng/ml) of TRIAC after a single topical administration, from baseline (hours) to 72 hours. | 0-72 hours
  MS-based method for analysis of TRIAC will be used.
Change in systemic levels (ng/ml) of DHEA-S after a single topical administration, from baseline (hours) to 72 hours. | 0-72 hours
  MS-based method for analysis of DHEA-S will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Roskilde University Hospital, Dept of Dermatology, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No